CLINICAL TRIAL: NCT05562362
Title: A Three Way Sequential, Randomised, Open-Label Study Designed to Evaluate the Single and Multiple-Dose Pharmacokinetics and the Effect of Food on the Single-Dose Pharmacokinetics of Oral Sparsentan Suspension in Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics of Oral Sparsentan Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTRX-RE021-102 (QSC200850)
Record Dates: First submitted 2022-08-23; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-06

CONDITIONS: Healthy Subjects
Keywords: Focal Segmental Glomerulosclerosis (FSGS); Immunoglobulin A Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Glomerulonephritis, IGA | interventions — sparsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fasted State (Experimental): Sparsentan will be administered in 3-dose level in healthy subjects. Subjects will be randomized to 1 of 3 dose levels (200mg, 400mg and 800 mg) and will receive a single dose of sparsentan in the fasted state on Period 1, Day 1 (Study Day 1)
  Interventions: Drug: RE-021, sparsentan
- Fed State (Experimental): Sparsentan will be administered in 3-dose level in healthy subjects. Subjects will have a single dose of sparsentan (200mg, 400mg and 800 mg) in the fed state (high-fat breakfast) on Period 2, Day 1 (Study Day 8)
  Interventions: Drug: RE-021, sparsentan
- Fed State - Multiple (Experimental): Sparsentan will be administered in 3-dose level in healthy subjects. Subjects will have multiple doses of sparsentan (200mg, 400mg and 800 mg) in the fed state on Period 3, Days 1 to 14 (Study days 12 to 25)
  Interventions: Drug: RE-021, sparsentan

INTERVENTIONS:
Drug: RE-021, sparsentan — RE-021, sparsentan - Subjects will be randomized 1 of 3 dose level

SUMMARY:
This single-center, open-label, randomized, single and multiple-dose, 3-way sequential study at 3 dose levels will be performed in healthy subjects. Subjects will be randomized to 1 of the 3 dose levels. In each dose level, subjects will be administered a single dose in the fasted state and then a single dose in the fed state, followed by 14 days of dosing to assess Pharmacokinetics (PK) following multiple dosing.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, single- and multiple-dose, 3-way sequential study at 3 dose levels in healthy subjects. For logistical purposes subjects will be admitted to the unit to be dosed in groups of approximately 16 or fewer. Subjects will be randomized into one of the three dose levels. Within each dose level, subjects will be administered a single dose in the fasted state and then a single dose in the fed state, followed by 14 days of dosing to assess PK following multiple dosing.

Subjects will undergo preliminary screening procedures for the study at the screening visit (Day -28 to Day -2). Subjects will be admitted to the clinical unit on the evening prior to investigational medicinal product (IMP) administration (Day -1) and will remain on site until 72 h post-final dose. Subjects will receive a single dose of sparsentan in the fasted state on Period 1, Day 1 (Study day 1) and a single dose of sparsentan in the fed state (high-fat breakfast) on Period 2, Day 1 (Study day 8), followed by multiple doses of sparsentan in the fed state on Period 3, Day 1 to 14 (Study days 12 to 25). On PK sampling days for the multiple dose treatment period (Period 3, Days 7, and 14; Study days 18 and 25), subjects will consume a high-fat breakfast before dosing; on other days, a standard breakfast will be provided.

A follow-up phone call will take place 5 to 7 days post-final dose to ensure the ongoing wellbeing of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or healthy females of non-childbearing potential
2. Between 18 and 55 years of age, inclusive, at time of signing informed consent
3. Body mass index (BMI) of 18.0 to 30.0 kg/m2 as measured at screening
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
2. Subjects who are or are immediate family members of a study site employee or a sponsor employee
3. Subjects who have previously been enrolled (dosed) in this study; subjects who have previously received sparsentan
4. Evidence current SARS-CoV-2 infection
5. History of any drug or alcohol abuse in the past 2 years
6. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
7. A confirmed positive alcohol breath test at screening or admission
8. Current smokers and those who have smoked within the last 3 months
9. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
10. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 3 months
11. Females of childbearing potential:

    * A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration ≥40 IU/L)
12. Subjects who are pregnant or lactating and subjects with pregnant or lactating partners. All women must have a negative pregnancy test at admission
13. Subjects who do not have suitable veins for multiple venipunctures/cannulation as assessed by the investigator or delegate at screening
14. Clinically significant abnormal clinical chemistry, hematology or urinalysis as judged by the investigator at screening
15. Serum alanine aminotransferase (ALT) > 1.5× upper limit of normal at screening
16. Serum potassium > upper limit of normal at screening
17. Confirmed positive drugs of abuse test result at screening or admission to Period 1
18. Corrected QT interval by Fridericia's formula (QTcF) greater than 450 msec; ventricular rate less than 40 per minute or greater than 90 per minute at screening or prior to dosing
19. For supine vital signs: systolic blood pressure less than 100 mmHg or greater than 140 mmHg (in subjects > 45 years of age up to 160 mmHg is acceptable); diastolic blood pressure less than 60 mmHg or over 90 mmHg at screening and pre-first dose.
20. Decrease in systolic blood pressure of 20 mmHg or more and/or decrease in diastolic blood pressure of 10 mmHg or more, measured after standing for approximately 2 to 5 min at screening and pre-dose in Period 1.
21. Increase in heart rate of over 30 bpm measured after standing for 2 to 5 min at screening and pre-dose Period 1
22. Any current or recent symptoms of postural hypotension or postural tachycardia at screening and pre-dose Period 1
23. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
24. Evidence of renal impairment at screening, as indicated by an eGFR of <90 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) (2009) equation
25. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
26. Subjects with a history of cholecystectomy or gall stones
27. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
28. Subjects with a history of any hypersensitivity to angiotensin receptor blockers, endothelin receptor antagonists or the suspension formulation excipients
29. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
30. Donation or loss of greater than 400 mL of blood within the previous 3 months
31. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than 4 g of paracetamol per day or hormone replacement therapy [HRT]) in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the PI
32. Use of any medication, eg erythromycin, itraconazole, and gestodene, that is known to inhibit CYP3A4 within 14 days before IMP administration
33. Use of any medication or substance known to induce CYP3A4, eg St John's Wort, within 30 days before IMP administration
34. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Assessment of single-dose pharmacokinetics of sparsentan oral suspension dosed in fed and fasted states - Cmax | Study Days 1 and 8
  Evaluation of, at minimum, the maximum concentration (Cmax) parameters for sparsentan following a single dose of sparsentan as an oral suspension in the fed or fasted state.
Assessment of single-dose pharmacokinetics of sparsentan oral suspension dosed in fed and fasted states - AUC(0-last) | Study Days 1 and 8
  Evaluation of, at minimum, the area under the concentration-time curve from dosing time 0 (AUC(0-last)) parameters for sparsentan following a single dose of sparsentan as an oral suspension in the fed or fasted state.
Assessment of single-dose pharmacokinetics of sparsentan oral suspension dosed in fed and fasted - states - AUC(0-inf) | Study Days 1 and 8
  Evaluation of, at minimum, the area under the concentration curve to infinite (AUC(0-inf)) time parameters for sparsentan following a single dose of sparsentan as an oral suspension in the fed or fasted state.
Food effect on pharmacokinetics of sparsentan oral suspension dosed after standard high-fat - breakfast - Cmax | Study Days 1 and 8
  Evaluation of the ratio, fed/fasted, for the Cmax
Food effect on pharmacokinetics of sparsentan oral suspension dosed after standard high-fat - breakfast - AUC(0-last) | Study Days 1 and 8
  Evaluation of the ratio, fed/fasted, for the AUC(0-last)
Food effect on pharmacokinetics of sparsentan oral suspension dosed after standard high-fat breakfast - AUC(0-inf) | Study Days 1 and 8
  Evaluation of the ratio, fed/fasted, for the AUC(0-inf)
Multiple-dose pharmacokinetics of a sparsentan oral suspension dosed in the fed state - Cmax | Study Days 12 to 28
  Evaluation of, at minimum, the following pharmacokinetics parameters for sparsentan following multiple doses of sparsentan as an oral suspension in the fed state: Cmax from a single dose for Study days 18 and 25 (Period 3, Days 7 and 14)
Multiple-dose pharmacokinetics of a sparsentan oral suspension dosed in the fed state - AUC(0-24) | Study Days 12 to 28
  Evaluation of, at minimum, the following pharmacokinetics parameters for sparsentan following multiple doses of sparsentan as an oral suspension in the fed state: Area under the plasma concentration-time curve over the last 24-h dosing interval (AUC(0-24)) from a single dose for Study days 18 and 25 (Period 3, Days 7 and 14)
Multiple-dose pharmacokinetics of a sparsentan oral suspension dosed in the fed state - TCP (AUC(0-24)/AUC(0-inf) | Study Days 12 to 28
  Evaluation of, at minimum, the following pharmacokinetics parameters for sparsentan following multiple doses of sparsentan as an oral suspension in the fed state: temporal change parameter (TCP) (AUC(0-24)/AUC(0-inf)) from a single dose for Study days 18 and 25 (Period 3, Days 7 and 14)

SECONDARY OUTCOMES:
Assessment of safety and tolerability of sparsentan oral suspension - clinical chemistry, hematology and eGFR | Study Days 1 to 28
  Safety laboratory tests including clinical chemistry, hematology and estimated glomerular filtration rate (eGFR) at each time point including virology and follicle stimulating hormone (FSH) (post-menopausal female subjects only) at screening
Assessment of Safety and tolerability of sparsentan oral suspension - vital sign (blood pressure) | Study Days 1 to 28
  Supine systolic and diastolic blood pressure (BP), including change from the baseline (Day 1, Pre-dose of each study period) will be summarized (ie, n -number of subjects with an observation, mean, SD - standard deviation, median, minimum and maximum) at each post-baseline time point by regimen. The number of subjects with 'substantial' increases or decreases or no substantial change from baseline in systolic BP (>20 mmHg), diastolic BP (>10 mmHg) will be summarized.
Assessment of Safety and tolerability of sparsentan oral suspension - vital sign (heart rate) | Study Days 1 to 28
  Supine heart rate, including change from the baseline (Day 1, Pre-dose of each study period) will be summarized (ie, n -number of subjects with an observation, mean, SD - standard deviation, median, minimum and maximum) at each post-baseline time point by regimen. The number of subjects with 'substantial' increases or decreases or no substantial change from baseline in heart rate (>15 bpm) will be summarized.
Assessment of Safety and tolerability of sparsentan oral suspension - ECG | Study Days 1 to 28
  Electrocardiogram (ECG) data, including change from baseline (Day 1, Pre-dose of each study period), will be summarized (ie, n -number of subjects with an observation, mean, SD - standard deviation, median, minimum and maximum)) at each post-baseline time point by regimen. The number and percentage of subjects with normal and prolonged QT intervals corrected for heart rate using Fridericia's correction (QTcF) and increases in QTcF intervals from baseline within the categories, defined as QTcF interval <=450 millisecond (msec), 451-480 msec, 481-500 msec, >500 msec, increase in QTcF interval from baseline <30 msec, 30-60 msec, >60 msec (based on the International Council on Harmonization [ICH] E14 guideline ) will be summarized at each post-baseline time point by regimen and time point.
Assessment of Safety and tolerability of sparsentan oral suspension - AEs | 2 to 28 days before Study Day 1 until 5 to 7 days post-final dose
  An AE is any untoward medical occurrence in a subject that occurs either before dosing (referred to as a pre-dose AE) or once a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product. Treatment-emergent adverse events (TEAEs) are AEs that commence during/after the first dose of investigational medicinal product (IMP) or commence before first dose of IMP (ie, a pre-dose AE or existing medical condition) but worsen in intensity during exposure to IMP. The number and percentage of subjects reporting each TEAE will be summarized for both System Organ Class (SOC) and Preferred Term (PT). For summaries by SOC and PT, with the exception of TEAEs by severity and relationship to IMP, the number of subjects and the number of events will be summarized. For summaries by severity and relationship only the number of subjects will be summarized.
Acceptability and key taste attributes of sparsentan oral suspension | Study Day 1
  Assess the palatability of the oral suspension using the results from a 9-point scale that rate acceptability of smell, sweetness, bitterness, flavor, mouth feel/texture, grittiness and aftertaste, and overall acceptability for a single dose of an oral suspension of sparsentan in the fasted state. Patient will rate overall liking of the product from a 9-point scale ranging from 1 = Dislike extremely and 9 = Like extremely.

CONTACTS AND LOCATIONS:
Locations (1):
- Travere Investigational Site, Nottingham, United Kingdom